CLINICAL TRIAL: NCT04880304
Title: Effects of Subconcussive Head Impacts on Neural Integrity and Function in ADHD: a Case-control Intervention
Brief Title: Effects of Subconcussive Head Impacts on Neural Integrity and Function in ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Assistant Professor Kinesiology, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2007515951
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Sport Injury; Attention-deficit/Hyperactivity Disorder
Keywords: Soccer Heading; Subconcussive Head Impacts; Attention-deficit/hyperactivity disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator who administers the semi-structured diagnostic interview for both groups using the Adult ADHD Investigator Symptom Rating Scale (AISRS), which is a robust, valid efficacy measure of ADHD symptoms in adult patients will be blinded to the study participants' diagnosis status. Additionally, the statistician will be blinded from group assignment. These processes will ensure single blind method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD diagnosis and subconcussive head impacts (Experimental): ADHD Group: Individuals clinically diagnosed with ADHD, currently taking his/her prescribed ADHD medication.
  Device: Soccer Heading Soccer Heading: Subjects stood approximately 40 feet away from a JUGS soccer ball launcher and participated in 20 consecutive soccer headings, separated by one minute intervals.
  Interventions: Other: Soccer Heading
- No history or current diagnosis of ADHD and subconcussive head impacts (Experimental): Non-ADHD Group: Individuals with no current or prior diagnosis of ADHD.
  Device: Soccer Heading Soccer Heading: Subjects stood approximately 40 feet away from a JUGS soccer ball launcher and participated in 20 consecutive soccer headings, separated by one minute intervals.
  Interventions: Other: Soccer Heading

INTERVENTIONS:
Other: Soccer Heading — A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer embedded in a head-band pocket and positioned directly below the external occipital protuberance (inion) to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 25mph. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practice and games. Subjects will stand approximately 40ft away from the machine to perform the heading. Participants perform 20 standing headers with 1 header per 30 seconds. The subjects will be instructed to direct the ball back toward the JUGS soccer machine in the air.
  Arms: ADHD diagnosis and subconcussive head impacts
Other: Soccer Heading — A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer embedded in a head-band pocket and positioned directly below the external occipital protuberance (inion) to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 25mph. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practice and games. Subjects will stand approximately 40ft away from the machine to perform the heading. Participants perform 20 standing headers with 1 header per 30 seconds. The subjects will be instructed to direct the ball back toward the JUGS soccer machine in the air.
  Arms: No history or current diagnosis of ADHD and subconcussive head impacts

SUMMARY:
The purpose of this study is to examine the acute neural responses to subconcussive head impacts in individuals with Attention-deficit/hyperactivity disorder (ADHD). The study is designed to identify the effects of 10 controlled soccer headings in college-aged soccer players diagnosed with ADHD and without ADHD, through the use of neural-injury blood biomarkers, functional and diffusion MRI, and ocular-motor function across three acute timepoints. The central hypothesis is that neuronal structural, physiological, and functional impairments from subconcussive head impacts will be amplified by ADHD. The neural-injury blood biomarkers neurofilament light (NF-L), glial fibrillary acidic protein (GFAP), ubiquitin C-terminal hydrolase-L1 (UCHL-1), and Tau will be measured in plasma, with the hypothesis that 10 soccer headings will significantly increase plasma NF-L levels in both groups at 24h post-heading compared to baseline, but this increase will be higher in the ADHD group; plasma UCH-L1, GFAP, and Tau levels will increase significantly after 10 headings in the ADHD group at 2h and 24h post-heading, but levels in the non-ADHD group will remain consistent throughout the time points. It is also hypothesized that repetitive subconcussive head impacts will impair neurocognitive function, as measured by regional changes in fMRI activation during working memory and attention-based tasks, in the ADHD group. Ten headings will significantly alter fMRI activation in the ADHD group from baseline. This impairment will not be observed in the non-ADHD group, rather the non-ADHD group will show consistent fMRI activation even after 10 headings. White matter microstructure will be measured by diffusion imaging metrics, with the hypothesis that 10 soccer headings will significantly disrupt microstructure in the ADHD group compared to baseline, but not in the non-ADHD group. The study will also assess neuro-ophthalmologic function as measured by the King-Devick test (KDT) and oculomotor function as measured by the near-point-of-convergence (NPC) in response to subconcussive head impacts. The hypothesis is that NPC performance will be significantly impaired and persist for longer than 24 hours in both groups, but this impairment will be greater in the ADHD group, and that the learning curve and expected improvement of KDT will be significantly blunted in both groups, with a display of worsening in the ADHD group.

DETAILED DESCRIPTION:
We will recruit participants on a first-come, first-served basis for the ADHD group. We will select age- and sex-matched controls (e.g., matched to 1st, 3rd, 5th, and 7th ADHD participants since this is 1:2 frequency-matched sampling) for the non-ADHD group. We propose to include a total of 60 participants in the study (ADHD n= 40, non-ADHD n=20).

The study consists of 3 data collection time points in a 2-day period. The 1st day will last approximately 4.75 hours and 2nd day will last approximately 1.5 hours. This study design will enable to test outcome measures over 2 acute phases.

* The 1st test session takes place right before the soccer heading intervention
* Participants will perform the soccer heading intervention
* The 2nd test session takes place 2 hours after the soccer heading intervention
* The 3rd test session takes place approximately 24 hours after the intervention

When written informed consent is obtained, we will use a self-reported health questionnaire to obtain demographic information. The information includes age, sex, BMI, race/ethnicity, years of soccer playing and heading experience, number and age of previous concussions, and sleep habits, as well as assessment of other neurological conditions to screen participants' eligibility. Participants who meet the inclusion criteria and are free of exclusionary factors will advance to the testing procedures. From 3 days before the study until the 24h post-heading time point, participants will be instructed to (1) take ADHD medication (for the ADHD Cohort), (2) refrain from consuming alcohol and recreational drugs, and (3) refrain from activities that involve head impacts.

Soccer Heading Intervention:

A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer and gyroscope (Triax Technologies) embedded in a head-band pocket and positioned back of the head to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 25mph across both groups. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practice and game. Participants will stand approximately 40ft away from the machine to perform soccer ball headings. An average linear head acceleration from a header sits around 20 g, while regular corner or goal kicks (~50mph) yield accelerations above 50 g. Participants in both groups will perform 10 headers with 1 header per minute.

Health Questionnaire Screening:

When written informed consent is obtained, we will use a self-reported health questionnaire to obtain demographic information. The information includes age, sex, BMI, race/ethnicity, years of soccer playing and heading experience, number and age of previous concussions, and sleep habits, as well as assessment of other neurological conditions to screen participants' eligibility. Before the first and final test session, participants will be asked to verify that they have slept longer than 4 hours the prior night, did not consume alcohol or recreational drugs within 3 days before the start of the study, did not participant in activities that involve head impacts within 3 days before the start of the study, and for the ADHD group they will be asked to provide the time of when they took their prescribed ADHD medication for the day. In addition, participants will complete a Participant Health Screening Checklist with the Imaging Research Facility (IRF) operator prior to participating in the imaging procedures. This checklist will screen participants for symptoms related to COVID-19.

ADHD Diagnosis and Screening of Psychiatric Factors and Substance Misuse:

We will use a two-step validation of ADHD diagnosis for both groups. Upon signing the consent form, ADHD participants will be instructed to submit confirmation of the ADHD diagnosis evaluated and assigned by their physicians. During a follow-up meeting, we will conduct a semi-structured diagnostic interview for both groups using the Adult ADHD Investigator Symptom Rating Scale (AISRS), which is a robust, valid efficacy measure of ADHD symptoms in adult patients. The assessment will be given by a trained examiner (a clinical social worker), who will be blinded from the participants' diagnosis status. We will also assess (1) depression, anxiety, and panic symptoms using the PHQ-9; (2) alcohol use disorder using AUDIT; and (3) cannabis use disorder using CUDIT.

NPC and KDT:

During each test session, various assessments will be conducted on each participant. First, ocular assessments consisting of near point of convergence (NPC) and the King-Devick Test (KDT) will be used to assed ocular-motor function and neuro-ophthalamolgic function, respectively. The NPC measures the closest point to which one can maintain convergence while focusing on an object before double vision occurs. Assessment will be repeated twice, and mean NPC scores will be used for statistical analyses. After they have finished NPC, participants will complete the KDT. The KDT assesses neuro-ophthalamogic function due to it's design of saccadic eye movements coupled with multiple facets of brain functions such as attention, language, and concentration. It will be administrated on a hand- held tablet. Participants will be given one trial "demonstration" card to practice the task. Following the demonstration card, participants will tap through 3 test cards. Participants will be asked to read aloud, left to right and top to bottom, a series of numbers on the test cards as fast and as accurate as they can while refraining from using his/her fingers as a reading guide. The 3 test cards progress in difficulty (i.e. guideline disappearance, numbers become more dense). The KDT records the total time, in seconds, participants spent to complete the task (all 3 test cards). Accuracy will be recorded by a lab personnel member who will stand behind the participant and record any errors (incorrect number, missed number, etc.) made during the testing.

Eye Reflex Assessment (Blinktbi):

The blink reflex is elicited when a stimulus is applied to or near the cornea, immediate area surrounding the canthus, the eyelashes, or directly to the peri-orbital nerves. This reflex is facilitated by stimulation to nerves that enter into the brainstem, loops through a number of brainstem and basal ganglia structures, including the reticular formation and the dopaminergic systems, and then out to the facial nerves as the actual blink. This provides a non-invasive way to monitor the integrity of the deep brain structures. It is postulated that by precisely measuring metrics associated with blink, data can be gathered on the field that will assist in detecting alterations in brain function suggestive of concussion or more severe brain injury. An FDA approved Eyestat device will be used for this testing.

Blood Biomarkers:

Antecubital vein blood draws will be performed each test session to help determine serum biomarker concentrations. A trained phlebotomist will thoroughly clean the inner elbow surface with an alcohol swab and draw 7 ml of whole blood into sterile Vacutainer tubes with 21G butterfly needle. After the blood draw, the participant will use gauze to maintain direct pressure and a bandage will be provided. Plasma will be assessed by the 4-plex Simoa assay platform (Quanterix), which is a magnetic bead-based ELISA that allows detection of biomarkers in femtomolar concentrations.

MRI Techniques:

Once completing the MRI screening procedure, participants will undergo the following standardized MRI protocols.

Diffusion tensor imaging (DTI) is the most widely used technique to study the microstructural integrity of white matter in vivo. DTI provides simple markers, such as mean diffusivity (MD) and fractional anisotropy (FA), that have been used to reflect microstructural tissue change during aging, neurological disorders, and traumatic brain injury (i.e., concussion). However, despite their sensitivity, MD and FA represent cellular diffusivity estimated by basic statistical descriptions that do not directly correspond to biophysiological parameters of the neural cellular integrity. DTI assumes Gaussian diffusion within a single microstructural compartment and thus has proven non-specific to axonal structural damage. To address this limitation, neurite orientation dispersion and density imaging (NODDI) has been characterized to assess microstructural integrity of axons using a non-Gaussian model with multiple compartments. NODDI allows researchers to measure axonal density within white matter, orientation of axonal dispersion, and free water diffusion. The combined approach using NODDI and DTI will uncover greater depth of progressive axonal degeneration in response to repetitive subconcussive head impacts.

Flanker Task: The Flanker test measures participants' ability to focus attention and ignore irrelevant information. Therefore, the Flanker task will assess the changes in attention in participants over time. For this task, while in the scanner, participants will be presented with a set of 5 arrows above the fixation point. They will be instructed to only respond to the direction of the central arrow. If the arrow is pointing to the left, participants will be instructed to press the index button of the controller in their left hand. If the arrow is pointing to the right, participants will be instructed to press the index button of the controller in their right hand. Participants will be read instructions prior to the test and will be permitted to press both index buttons to assure there is an understanding. The task will run for a total of approximately 10 minutes.

N-Back Tasks: The n-back task will be used to asses both verbal (letters) and visual (blocks) memory. For the verbal n-back tasks, while in the scanner, participants will be presented a series of letters, with letters being displayed on the screen one at a time. Participants will be instructed to answer whether the target letter is the same or different from the letter presented, if it the presented target is the same or different from the letter presented 1-back or 2-back letters prior. If the target letter is the same, participants will be instructed to press the index button of the controller in their left hand and if the letter is different, participants will be instructed to press the index button of the controller in their right hand. For the visual n-back tasks, the design and instructions will be the same, but letters will be replaced with simple abstract objects. Participants will be read instructions prior to the test and will be permitted to press both index buttons to assure there is an understanding. The n-back tasks are performed as a block design, with a total duration of about 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

For ADHD Cohort

1. Aged between 18 and 26 years at the start of the study
2. Providing documentation of ADHD being clinically diagnosed by a psychologist, psychiatrist, or a neurologist 3) Taking their prescribed ADHD medication >5 days a week

4) Currently playing soccer (i.e., intercollegiate, intramural, club) 5) At least 5 years of soccer heading experience

For non-ADHD Cohort

1. Aged between 18 and 26 years at the start of the study
2. Absence of prior or current clinical diagnoses of ADHD
3. Absence of prior or current history of taking ADHD medication 4) Currently playing soccer (i.e., intercollegiate, intramural, club) 5) At least 5 years of soccer heading experience

Exclusion Criteria:

For both ADHD and non-ADHD Cohorts

1. Any head or neck injury in the year before the start of the study
2. Current use of medications that trigger drowsiness
3. Pregnancy
4. Any history of neurological disorders and learning disability other than ADHD
5. Metal implants in the head
6. Implanted electro/magnetic devices (e.g. orthodontic braces, pacemakers, aneurysm clips)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Acute change in brain-derived blood biomarkers from pre to 2 hour post-heading | Blood samples will be collected at pre- and 2 hour post-heading
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), tau, and Ubiquitin C-terminal Hydrolase 1 (UCH-L1). All expression levels in pg/mL.
Acute change in brain-derived blood biomarkers from pre to 24 hour post-heading | Blood samples will be collected at pre- and 24 hour post-heading
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum samples will be assayed for neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), tau, and Ubiquitin C-terminal Hydrolase 1 (UCH-L1). All expression levels in pg/mL.
Acute change in regional fMRI activation during memory and attention tasks from pre to 2 hour post-heading | fMRI procedures will be performed at pre and 2 hour post-heading
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with an eight channel phased array head radiofrequency coil will be used to collect fMRI images while attention and working memory tasks are administered.
  The task based fMRI protocol will consist of N-Back tasks to assess visual and verbal working memory, Flanker task to assess attention, and a function Resting State task.
Acute change in regional fMRI activation during memory and attention tasks from pre to 24 hour post-heading | fMRI procedures will be performed at pre and 2 hour post-heading
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with an eight channel phased array head radiofrequency coil will be used to collect fMRI images while attention and working memory tasks are administered.
  The task based fMRI protocol will consist of N-Back tasks to assess visual and verbal working memory, Flanker task to assess attention, and a function Resting State task.
Acute change in axonal microstructure from pre to 2 hour post-heading. | MRI procedures will be performed at pre and 2 hour post-heading
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with an eight channel phased array head radiofrequency coil will be used to assess changes in diffusion metrics.
  Whole-brain Diffusion tensor imaging (DTI) will be performed with a multi-slice single-shot spin echo echoplanar pulse sequence (echo time [TE] = 81 ms; repetition time [TR] = 9 s) using 64 diffusion-encoding directions, isotopically distributed over the surface of a sphere with electrostatic repulsion.
  Neurite orientation, dispersion and density imaging (NODDI) metrics will be used in addition to DTI to assess axonal density within white matter, orientation of axonal dispersion, and free water diffusion.
Acute change in axonal microstructure from pre to 24 hour post-heading. | MRI procedures will be performed at pre and 24 hour post-heading
  A standardized MRI protocol acquired on a Siemens TIM Trio scanner, equipped with an eight channel phased array head radiofrequency coil will be used to assess changes in diffusion metrics.
  Whole-brain Diffusion tensor imaging (DTI) will be performed with a multi-slice single-shot spin echo echoplanar pulse sequence (echo time [TE] = 81 ms; repetition time [TR] = 9 s) using 64 diffusion-encoding directions, isotopically distributed over the surface of a sphere with electrostatic repulsion.
  Neurite orientation, dispersion and density imaging (NODDI) metrics will be used in addition to DTI to assess axonal density within white matter, orientation of axonal dispersion, and free water diffusion.

SECONDARY OUTCOMES:
Acute change in ocular-motor function from pre to 2 hour post-heading | Ocular-motor function will be assessed at pre- and 2 hour post-heading
  Participants will undergo 3 ocular-motor assessments: 1) near-point of convergence; 2) King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing; and 3) Blinktbi--a blink reflex assessment.
Acute change in ocular-motor function from pre to 24 hour post-heading | Ocular-motor function will be assessed at pre- and 24 hour post-heading
  Participants will undergo 3 ocular-motor assessments: 1) near-point of convergence; 2) King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing; and 3) Blinktbi--a blink reflex assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be included in publications.

REFERENCES:
- [Background] Biederman J, Feinberg L, Chan J, Adeyemo BO, Woodworth KY, Panis W, McGrath N, Bhatnagar S, Spencer TJ, Uchida M, Kenworthy T, Grossman R, Zafonte R, Faraone SV. Mild Traumatic Brain Injury and Attention-Deficit Hyperactivity Disorder in Young Student Athletes. J Nerv Ment Dis. 2015 Nov;203(11):813-9. doi: 10.1097/NMD.0000000000000375. PMID 26461480
- [Background] Iaccarino MA, Fitzgerald M, Pulli A, Woodworth KY, Spencer TJ, Zafonte R, Biederman J. Sport concussion and attention deficit hyperactivity disorder in student athletes: A cohort study. Neurol Clin Pract. 2018 Oct;8(5):403-411. doi: 10.1212/CPJ.0000000000000525. PMID 30564494
- [Background] Nowak MK, Bevilacqua ZW, Ejima K, Huibregtse ME, Chen Z, Mickleborough TD, Newman SD, Kawata K. Neuro-Ophthalmologic Response to Repetitive Subconcussive Head Impacts: A Randomized Clinical Trial. JAMA Ophthalmol. 2020 Apr 1;138(4):350-357. doi: 10.1001/jamaophthalmol.2019.6128. PMID 32053162
- [Background] Wirsching A, Chen Z, Bevilacqua ZW, Huibregtse ME, Kawata K. Association of Acute Increase in Plasma Neurofilament Light with Repetitive Subconcussive Head Impacts: A Pilot Randomized Control Trial. J Neurotrauma. 2019 Feb 15;36(4):548-553. doi: 10.1089/neu.2018.5836. Epub 2018 Sep 4. PMID 30019617
- [Derived] Nowak MK, Kronenberger WG, Rettke D, Ogbeide O, Klemsz LM, Quinn PD, Mickleborough TD, Newman SD, Kawata K. Neuro-ophthalmologic and blood biomarker responses in ADHD following subconcussive head impacts: a case-control trial. Front Psychiatry. 2023 Nov 22;14:1230463. doi: 10.3389/fpsyt.2023.1230463. eCollection 2023. PMID 38076682